CLINICAL TRIAL: NCT06371573
Title: Ultrasound Examination for Spleen Volume Evaluation in Myeloproliferative Neoplasms: Comparison With MRI Examination
Brief Title: Ultrasound Examination for Spleen Volume Evaluation in Myeloproliferative Neoplasms
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Full Professor, Federico II University
Other Study IDs: MPN-USspleen
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Myeloproliferative Neoplasm; Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis; Prefibrotic/Early Primary Myelofibrosis
Keywords: Ultrasound; MRI; Myeloproliferative Neoplasm; Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis; Prefibrotic/Early Primary Myelofibrosis; spleen
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ULTRASOUND EXAM AND MRI SCAN — Within two weeks from the US, each patient underwent an MRI of the upper abdomen to evaluate the splenic volume. MRI examinations were performed using a 3T Biograph mMR scanner (Siemens Healthcare, Erlangen, Germany) with 4-channel flex phased-array body coil. Routine clinical abdominal MRI acquisition includes coronal T2W Half-Fourier Acquisition Single-shot Turbo spin Echo imaging (HASTE), axial T1 Dual-echo FSE, axial T2 TSE Fat Sat, and an axial diffusion-weighted imaging (DWI).

SUMMARY:
Adult patients (>18 years) with newly diagnosis of Ph negative myeloproliferative neoplasms (MPNs) according to WHO 2016 criteria, will be recruited to this study.

This study is the result of the collaboration the Hematology Division of Federico II University Medical School of Naples (Italy), that performed the US investigation and the IRCCS SYNLAB SDN where the patients carried out MR. The study is conducted in accordance with the Declaration of Helsinki. All subjects gave informed consent to receive both US and MR scans of the spleen.

All spleen US scans were performed by the same operator (with>10 years of experience in abdominal US), who used an EPIQ 5 Philips instrument with a 1-5 MHz broadband curvilinear probe. The spleen was scanned in patients who were fasting, in the longitudinal and transverse planes by using an intercostal approach, a subcostal approach, or both.

The patient was placed in a supine or right-sided position until complete organ visualization was achieved. Perimeter, longitudinal diameter (LD), and area, defined as the maximum measurements with splenic borders and angles clearly defined, were measured, and SV (in milliliters) was calculated automatically. For each subject, the mean value of 3 measurements repeated on the same imaging session was calculated and recorded for final analysis. Within two weeks from the US, each patient underwent an MRI of the upper abdomen to evaluate the splenic volume. MRI examinations were performed using a 3T Biograph mMR scanner (Siemens Healthcare, Erlangen, Germany) with 4-channel flex phased-array body coil. Routine clinical abdominal MRI acquisition includes coronal T2W Half-Fourier Acquisition Single-shot Turbo spin Echo imaging (HASTE), axial T1 Dual-echo FSE, axial T2 TSE Fat Sat, and an axial diffusion-weighted imaging (DWI). The DWI includes an apparent diffusion coefficient (ADC) map that was automatically generated at the time of acquisition. At last, an isotropic 2mm3 axial Volumetric Interpolated Breath-hold Examination (VIBE) sequence for SV evaluation was acquired. For the latter, attention was paid to optimize the field of view to the spleen, in order to reduce patient's apnea and possible respiratory artifacts. A radiologist with mote than 10 years of experience in abdominal MRI reporting performed measurement of the three orthogonal diameters of the spleen for each patient. Subsequently, SV was calculated using ITK-SNAP software and semi-automatic 3D segmentation approach, firstly based on a signal threshold.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Philadelphia (Ph) negative chronic myeloproliferative neoplasms (MPN), according to WHO 2016 criteria
* age >18 years
* execution of MRI of the upper abdomen within two weeks from the US,

Exclusion Criteria:

* patients not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, non-interventional study. Data were retrospectively collected from all patients who completed US and MRI scans
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
agreement between two different diagnostic methods | 2 weeks
  Estimation of Spleen Volume and Longitudinal Diameter obtained with US measurement were compared to that obtained using MRI conducted in a time span of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No